CLINICAL TRIAL: NCT02449603
Title: Comparison of Exenatide vs. Biphasic Insulin Aspart 30 on Glucose Variability in Type 2 Diabetes : a Randomised Open Parallel-controlled Study
Brief Title: Comparison of Exenatide vs. Biphasic Insulin Aspart 30 on Glucose Variability in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other); Chang'An Hospital (Other); Xi'an Gaoxin Hospital (Other); Xi'an Central Hospital (Other); Shaanxi Aerospace Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10319
Record Dates: First submitted 2015-05-11; First posted 2015-05-20 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Chinese population
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): Exenatide (Colorless transparent liquid, comes in a prefilled pen.5ug/10ug, AstraZeneca) should be initiated, 60 minutes pre-breakfast and pre-supper, at 5ug twice a day for 4 weeks and then titrated up at 10ug twice a day until the completion of the study.
  Interventions: Drug: Exenatide
- Biphasic insulin Aspart 30 (Active Comparator): Biphasic insulin Aspart 30 (Colorless transparent liquid, 100u/mL, 3ml each, Novo Nordisk), subcutaneous injection, starting at a dose of 0.2-0.4 IU/kg, or 10～12 IU/d assigned in pre-breakfast and pre-supper in a 1:1 ratio. The adjustment of insulin dose is instructed to achieve an optimal balance between glycaemic control and risk of hypoglycaemia as dictated by best clinical practice, titrated to glucose targets of fasting plasma glucose (FPG) and pre-supper <7 mmol/L.
  Interventions: Drug: Biphasic insulin Aspart 30

INTERVENTIONS:
Drug: Exenatide
  Other Names: Byetta
  Arms: Exenatide
Drug: Biphasic insulin Aspart 30
  Arms: Biphasic insulin Aspart 30

SUMMARY:
This is a multi-centre, open-label, randomized, parallel trial to compare the effect of Exenatide versus Biphasic insulin Aspart 30 on glucose variability and inflammatory markers in type 2 diabetes mellitus (T2DM) patients inadequately controlled with metformin monotherapy.

DETAILED DESCRIPTION:
Studies have showed that fluctuations of glucose seem to have more deleterious effects than sustained hyperglycaemia in the development of diabetic complications. The present randomized controlled trial was designed with primary aim to evaluate glycaemic fluctuation in the comparison between twice-daily Exenatide and other treatment paradigm (e.g. insulin Aspart 30).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Men and women (non-pregnant and using a medically approved birth-control method) aged between 18 and 70 years at screening.
* Confirmed type 2 diabetes with history of at least half a year.
* Treatment with stable, maximum tolerated doses of metformin (≧1500mg/d, ≧3 months).
* HbA1c ≥ 7.5% and ≤ 10.0% at screening or within 4 weeks prior to screening (by local laboratory).
* Body mass index: 21-35 kg/m^2.

Exclusion Criteria:

* Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.
* Diagnosis or history of:

  1. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury or secondary forms of diabetes, e.g., acromegaly or Cushing's syndrome.
  2. Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months.
* Previous treatment with any dipeptide peptidase-4 (DPP4) inhibitor or glucagon-like peptide-1 (GLP-1) receptor agonists within the past one year.
* History of hypersensitivity reaction (e.g., anaphylaxis, angioedema, exfoliative skin conditions) to dipeptide peptidase-4 inhibitor (DPP4) or Acarbose.
* Treatment with any anti-diabetic medication for more than 7 consecutive days other than metformin in the last 3months prior to screening.
* Treatment with systemic glucocorticoids (oral, intravenous) for more than consecutive 7 days within the past 6 months.
* Triglycerides (fasting) > 4.5 mmol/L (> 400 mg/dL) at screening or within 4 weeks prior to screening (by local laboratory).
* Patients with clinically apparent liver disease characterized by either one of the following:

  1. Alanine transaminase (ALT) or aspartate aminotransferase (AST) > 3x upper limit of normal (ULN) confirmed on two consecutive measurements (by local laboratory) within 4 weeks prior to screening period
  2. Impaired excretory (e.g. hyperbilirubinemia) and/or synthetic function, or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites and bleeding from oesophageal varices.
  3. Acute viral or active autoimmune, alcoholic, or other types of hepatitis.
* Patients with moderate /severe renal impairment or end-stage renal disease (estimated Glomerular Filtration Rate ≤ 60 mL/min calculated by using the abbreviated equation developed by the Modification of Diet in Renal Disease (MDRD) study with modification for the Chinese population) at screening or within 4 weeks prior to screening (by local laboratory)
* Congestive heart failure defined as New York Heart Association (NYHA) class III or IV.
* Significant cardiovascular history within the past 3 months prior to screening defined as: myocardial infarction, coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident.
* History of chronic pancreatitis or idiopathic acute pancreatitis.
* History of gastrointestinal disease including gastroenterostomy, enterectomy, Roemheld Syndrome, severe hernia, intestinal obstruction, intestinal ulcer.
* History of genetic galactose intolerance, Lapp lactase deficiency and glucose-galactose malabsorption.
* History of medullary thyroid carcinoma.
* Diagnosed and/or treated malignancy (except for basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) within the past 5 years.
* History of organ transplant or acquired immunodeficiency syndrome (AIDS).
* History of alcohol abuse or illegal drug abuse within the past 12 months.
* Potentially unreliable patients and those judged by the Investigator to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change of mean amplitude of glycemic excursions | from baseline to Week 16

SECONDARY OUTCOMES:
HbA1c | at baseline and Week 16
Hours of hypoglycemia as measured by continuous glucose monitoring system (CGMS) | at baseline and Week 16
Blood pressure | at baseline and Week 16
Lipids | at baseline and Week 16
Body mass index | at baseline and Week 16
Waist circumference | at baseline and Week 16
Monocyte chemotactic protein-1 (MCP-1) | at baseline and Week 16
High-sensitivity C-reactive protein (hs-CRP) | at baseline and Week 16
Urinary albumin | at baseline and Week 16
Number of participants with adverse events/severe adverse events | from baseline to Week 16
Number of participants with clinical hypoglycemia | from baseline to Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Fourth Military Medical university, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wang L, Liu X, Yang W, Lai J, Yu X, Liu J, Gao X, Ming J, Ma K, Xu J, Tian Z, He Q, Ji Q. Comparison of Blood Glucose Variability Between Exenatide and Biphasic Insulin Aspart 30 in Chinese Participants with Type 2 Diabetes Inadequately Controlled with Metformin Monotherapy: A Multicenter, Open-Label, Randomized Trial. Diabetes Ther. 2020 Oct;11(10):2313-2328. doi: 10.1007/s13300-020-00904-z. Epub 2020 Aug 27. PMID 32856226
- [Derived] Xu S, Liu X, Ming J, Ji Q. Comparison of exenatide with biphasic insulin aspart 30 on glucose variability in type 2 diabetes: study protocol for a randomized controlled trial. Trials. 2016 Mar 24;17:160. doi: 10.1186/s13063-016-1258-8. PMID 27009108